CLINICAL TRIAL: NCT04017871
Title: Evaluation of Functional, Neuroplastic and Biomechanical Changes Induced by an Intensive, Playful Early-morning Treatment Including Lower Limbs (EARLY-HABIT-ILE) in Preschool Children With Uni and Bilateral Cerebral Palsy
Acronym: HABIT-ILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Fondation Paralysie Cérébrale (Other); Université Catholique de Louvain (Other); University of Pisa (Other); University of Lausanne Hospitals (Other); University Angers (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EARLY_HABIT-ILE (29BRC19.0050)
Record Dates: First submitted 2019-05-10; First posted 2019-07-12 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy (CP); pre-school children with unilateral and bilateral CP
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): 10 days of intensive and structured motor therapy, 5 hours a day = 50h
  Interventions: Other: MRI; Other: Electro-Encephalography-High Density (children with unilateral PC only); Other: 3D and EMG analysis; Other: care and classic activities; Device: Accelerometers
- Control (Placebo Comparator): 10 days of care and classic activities
  Interventions: Other: MRI; Other: Electro-Encephalography-High Density (children with unilateral PC only); Other: 3D and EMG analysis; Other: care and classic activities; Device: Accelerometers

INTERVENTIONS:
Other: MRI — MRI at baseline and J90
Other: Electro-Encephalography-High Density (children with unilateral PC only) — Electro-Encephalography-High Density (children with unilateral PC only) at baseline and J90
Other: 3D and EMG analysis — 3D and EMG analysis at baseline and J90
Other: care and classic activities — physiotherapy and psychomotility. As needed weekly sessions of speech therapist or orthoptist and daily activities of the child.
Device: Accelerometers — During 5 days a sensor at each wrist to quantify their movement.

SUMMARY:
An urgent priority in the field of paediatric neurorehabilitation is the development of effective early motor interventions.

Hand and Arm Bimanual Intensive Therapy Including Lower Extremities (= HABIT-ILE) applies the concepts of motor skill learning and intensive training to both the Upper Extremities (UE) and Lower Extremities (LE) and has been shown to improve aspects of motor function of the UE and LE in school age children with unilateral and bilateral Cerebral Palsy (CP) across the 3 levels of the International Classification of Functioning, Disability and Health (ICFDH). The principles and content of HABIT-ILE can be applied to pre-school children and this method is highly promising for early rehabilitation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of two weeks of early HABIT-ILE on gross motor function in pre-school children with unilateral and and bilateral Cerebral Paralysy (CP), in comparison with two weeks of usual motor activity including usual rehabilitation (control group).

ELIGIBILITY:
Inclusion Criteria:

* Child with unilateral cerebral palsy or Child with bilateral cerebral palsy proven spastic or dyskinetic
* Aged from 1 to 4 years old (12 to 59 months) (age corrected if prematurity) able to follow instructions and to be able to carry out all the evaluations, according to his age

Exclusion Criteria:

* Age> 2 years old (35 months) or 4 years old (59 months) during the internship evaluation period
* Uncontrolled epilepsy
* History of botulinum toxin injection or surgery in the 6 months preceding the study period or scheduled within 3 months (during the study period)
* Visual or cognitive impairment that may interfere with the management
* Common contraindications to magnetic resonance imaging (MRI) such as metal implants

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Assistive Hand Assesment (AHA/miniAHA) (for unilateral CP only) | 1 hour
  measures and describes how children with upper limb disability in one hand use his/her affected hand collaboratively with the non affected hand in bimanual play.The score range from 0 to 100 as a percentage. 100 is the best outcome.
Gross Motor Function Measure (GMFM) (for bilateral CP only) | 1 hour
  measures change in gross motor function over time in children with cerebral palsy. The score range from 0 to 100 as a percentage. 100 is the best outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Les Capucins, Angers
  - Fondation ILDYS - Site de Ty Yann, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Araneda R, Sizonenko SV, Newman CJ, Dinomais M, Le Gal G, Ebner-Karestinos D, Paradis J, Klocker A, Saussez G, Demas J, Bailly R, Bouvier S, Nowak E, Guzzetta A, Riquelme I, Brochard S, Bleyenheuft Y. Protocol of changes induced by early Hand-Arm Bimanual Intensive Therapy Including Lower Extremities (e-HABIT-ILE) in pre-school children with bilateral cerebral palsy: a multisite randomized controlled trial. BMC Neurol. 2020 Jun 12;20(1):243. doi: 10.1186/s12883-020-01820-2. PMID 32532249